CLINICAL TRIAL: NCT04898036
Title: Phototherapy For Treatment Of Raynaud's Phenomenon
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding or staff
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RHEUM-2021-29567
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Raynaud Disease; Raynaud Phenomenon; Raynaud Syndrome
MeSH Terms: conditions — Raynaud Disease | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham First, then Experimental (Experimental): Participants in this group will receive the sham treatment first, then the experimental treatment.
  Interventions: Device: Blue Light Therapy; Device: Sham Light Therapy
- Experimental First, then Sham (Experimental): Participants in this group will receive the experimental treatment first, then the sham treatment.
  Interventions: Device: Blue Light Therapy; Device: Sham Light Therapy

INTERVENTIONS:
Device: Blue Light Therapy — This phototherapy device (PTD-1) consists of a Plexiglas hand compartment (cleanable) enclosed in a powder-coated steel cabinet. Within the cabinet are two blue LED panels located above and below the hand compartment to illuminate the hands.
Device: Sham Light Therapy — To turn the device into a sham mode, a thin opaque liner can be inserted which will block light from illuminating the hands.

SUMMARY:
To determine if blue light therapy can improve the symptoms of Raynaud's phenomenon, and provide parameters for ultimately designing commercial treatment devices, an investigational stationary phototherapy unit was designed and built.

DETAILED DESCRIPTION:
The purpose of this study is to test the efficacy of blue light phototherapy for the treatment of Raynaud's phenomenon (RP) in human participants. The specific aim is to see if phototherapy treatment applied to the hands will reduce the symptoms that RP participants experience. This will be measured through the use of a visual analog scale (VAS) of both pain and numbness. This study will also help to infer whether blue light phototherapy causes vasodilation through infrared thermal imaging of the hands and continuous measurement of skin temperature with a surface thermistor. Together, the visual analog scale (VAS) and infrared thermal imaging contribute to the objective of deducing whether blue light phototherapy can lead to reduced RP symptoms due to vasodilation of blood vessels.

ELIGIBILITY:
Inclusion Criteria:

- Must have a current diagnosis by a physician of Raynaud's Phenomenon/Syndrome

Exclusion Criteria:

* Those with active ischemic digital ulcers or gangrene as the cold exposure can be a safety hazard for them.
* Inability of the subject to place their hands into the PTD portal because of physical size or discomfort.
* Inability of the subject to wear protective eyewear.
* Anyone, who in the judgement of any of the investigators, would be unable to safely complete the study procedures.
* Females who are pregnant.
* Adults unable to consent for any reason not explicitly stated herein.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) of Pain | 4 hours
  Participants will be asked to rate their pain upon cold room exposure between treatments using a 10 centimeter visual analog scale (VAS). Outcome is reported as the mean change in VAS per arm in units of millimeters.
Change in Visual Analog Scale (VAS) of Numbness | 4 hours
  Participants will be asked to rate their numbness upon cold room exposure between treatments using a 10 centimeter visual analog scale (VAS). Outcome is reported as the mean change in VAS per arm in units of millimeters.

SECONDARY OUTCOMES:
Skin Temperature | 4 hours
  Skin temperature of at least one finger will be measured and logged using a thermometer at multiple points during study visit. Outcome is reported in units of degrees Celsius.

OTHER OUTCOMES:
Thermal Imaging | 4 hours
  The thermal imaging camera takes still images of the hand before and immediately after treatment. It provides a heat map (color contour) that may be probed afterwards for temperature at designated points. These points are distributed over the fingers, hand and palms. A technician manually reads the temperature in degrees Celsius and enters the values into an Excel spreadsheet designating subject, ID and date; location of measurement; and other temperature readings. These include ambient (room temperature), and outside temperature. The finger and room temperatures, in Celsius, are electronically recorded on an Omega data logger. This is interrogated later to retrieve data. Another continuous reading is obtained of the temperature inside the hand compartment (separate from internal thermoregulation measurements) to track equipment functionality.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Molitor, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided